CLINICAL TRIAL: NCT07344324
Title: A Pilot Study Evaluating the Safety, Feasibility, and Therapeutic Potential of Endoscopic Duodenal Injection of Adipose Tissue-Derived Mesenchymal Stem Cells in Patients With Type 2 Diabetes Mellitus.
Brief Title: Study Evaluating the Safety and Feasibility of Endoscopic Duodenal Injections of Autologous Mesenchymal Stem Cells
Acronym: STEM-DM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7976
Record Dates: First submitted 2025-12-22; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: Diabete Type 2; Insulin Resistant Diabetes (Mellitus); Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 15 participants with T2DM (Experimental): Subjects with a BMI between ≥ 25 and ≤ 35 kg/m2, T2DM and age between 30-65 will be considered eligible for the study.
  Interventions: Procedure: endoscopic duodenal injection of ADMSCs

INTERVENTIONS:
Procedure: endoscopic duodenal injection of ADMSCs — Biopsy Protocol Mucosal biopsies (12 at baseline; 6 at follow-up) will be collected from the Treitz angle to the genu inferius. Samples for ex vivo analysis will be transported at 37°C in sterile medium within 15 minutes.
  ADMSC Preparation and Delivery Autologous adipose tissue, harvested via mini-liposuction, will undergo mechanical activation (ELEA Method: 2000 rpm for 8 min). The activated fat is filtered (2 mm), emulsified, and loaded into a 19-gauge needle. Under deep sedation, the substrate will be injected submucosally from the Treitz angle to the superior duodenal genu, ensuring papilla preservation.

SUMMARY:
Type 2 Diabetes Mellitus (T2DM) pathogenesis increasingly involves "diabetic duodenopathy," characterized by proximal intestinal immune and epithelial dysregulation. This study investigates the endoscopic delivery of adipose-derived mesenchymal stem cells (ADMSCs) into the duodenum and proximal jejunum as a disease-modifying therapy. By leveraging the paracrine immunomodulatory and regenerative effects of ADMSCs in close proximity to the pancreatico-enteroendocrine system, this targeted approach aims to restore insulin sensitivity and $\beta$-cell function while minimizing systemic exposure. The clinical safety and feasibility of this novel delivery route remain to be established.

ELIGIBILITY:
Inclusion Criteria:

* • Adults aged between 25-70 years

  * Diagnosis of T2DM from at least 1 years
  * HbA1c between 7.5% and 10%
  * BMI between 25 and 35 kg/m²
  * Fasting C-peptide ≥1 ng/ml
  * Stable antidiabetic regimen for ≥3 months (including insulin s.c.)
  * Insulin resistance (HOMA-IR > 5)
  * Healthy volunteers: BMI < 25, age between 18-75 and no diagnosis of T2DM or insulin resistance (HOMA-IR<2.5), with no significant acute or chronic medical conditions and not taking medications that could interfere with the esophagogastroduodenoscopy + biopsies

Exclusion Criteria:

* Type 1 DM or secondary diabetes
* Celiac disease
* History of pancreatitis or GI surgery
* Active infection or malignancies ongoing
* Active gastro-duodenal ulcers
* Duodenum not accessible endoscopically for previous surgery or other conditions
* History of autoimmune disease
* Active malignancy or recent cancer treatment
* Use of certain medications (e.g., immunosuppressants, systemic corticosteroids)
* Active Smoking (>5 sigarettes/die)
* Anticoagulant treatment not suspendable
* Myocardial infarction during the past 6 months or/and heart failure class III or IV according to the New York Heart association's classification.
* Drug or alcohol abuse
* Continuous glucocorticoid or anti-inflammatory treatment
* Uncontrolled thyroid disease.
* Pregnancy, breastfeeding
* Psychiatric or cooperative problems or low compliance that is a contraindication from participating in the study.
* Liver cirrhosis of any Child-Phugh stage or MELD> 15
* Chronic Severe Renal Insufficiency (eGFR < 30 ml/min/1.73 m2 based on CKD-EPI equation)
* Currently participating in other study, or previously participated in an experimental drugs trial within 30 days before or 5 half-life of the drug administered
* Any health issue that might put the patient at risk if the treatment is performed, judged by the investigator.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2027-02-02 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Related Adverse Events as Assessed by Common Terminology Criteria for Adverse Events Version 5.0 | From the time of the endoscopic procedure through Month 12 post-procedure.
  Assessment of the safety and tolerability of the endoscopic duodenal injection of autologous adipose tissue-derived Mesenchymal Stem Cells. Safety will be evaluated by monitoring the frequency and severity of all adverse events and serious adverse events occurring during the study period.

SECONDARY OUTCOMES:
Change From Baseline in Glycated Hemoglobin at Month 12 | Baseline (Day 0) and Month 12.
  Mean change from baseline in Glycated Hemoglobin (HbA1c) levels. This physiological parameter is used to evaluate the long-term control of blood sugar levels. The data will be aggregated as the mean change from the start of the study to the final follow-up.
Change From Baseline in Total Daily Insulin Requirement at Month 12 | Baseline (Day 0) and Month 12.
  Mean change from baseline in the total daily dose of insulin required by the participant. The dose is measured in International Units per Kilogram per Day. This measure assesses if the treatment reduces the patient's dependence on external insulin.
Change From Baseline in Fasting C-peptide Levels at Month 12 | Baseline (Day 0) and Month 12.
  Mean change from baseline in fasting C-peptide levels. This parameter is used as a surrogate marker for endogenous insulin production and pancreatic beta-cell function. It is measured in nanograms per milliliter.
Change From Baseline in Lipid Profile Parameters at Month 12 | Baseline (Day 0) and Month 12.
  Mean change from baseline in lipid profile parameters, including Total Cholesterol, Low-Density Lipoprotein (LDL), High-Density Lipoprotein (HDL), and Triglycerides. These physiological parameters are measured in milligrams per deciliter (mg/dL) to evaluate the metabolic impact of the Mesenchymal Stem Cell transplantation. Data will be aggregated as the mean change for each lipid component.

CONTACTS AND LOCATIONS:
Overall Officials: IVO BOSKOSKI, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS